CLINICAL TRIAL: NCT05871203
Title: Changes in Gene Expression and Prognosis of Blood Immune Cells After Cardiopulmonary Bypass Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0359
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Cardiopulmonary bypass; gene expression
MeSH Terms: conditions — Acute Kidney Injury | interventions — Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative acute kidney injury
  Interventions: Other: Gene sequencing
- Postoperative non-acute kidney injury
  Interventions: Other: Gene sequencing

INTERVENTIONS:
Other: Gene sequencing — Participants were taken blood samples for gene sequencing at three time periods: before, after, and 24 hours after the end of the surgery

SUMMARY:
The goal of this observational study is to learn about the changes in gene expression in blood immune cells in after cardiac surgery with cardiopulmonary bypass.The main question it aims to answer is: What specific gene expression changes predict kidney damage after cardiac surgery with cardiopulmonary bypass. Participants received conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age≥ 18 years old; 2) Cardiopulmonary bypass descending valve replacement (molding), or coronary artery bypass grafting, or macrovascular surgery.

Exclusion Criteria:

* 1) any cognitive or mental impairment that is unable to sign the informed consent form; 2) Have basic immune system and blood system diseases; 3) pregnancy; 4) Receiving radiotherapy and chemotherapy before surgery; 5) Receiving immunosuppressive drugs within six months; 6) Have participated in other interventional clinical trials within 30 days before surgery.

Exit Criteria:

1. Incomplete surgery;
2. Secondary transfer in the operating room;
3. Automatically request to terminate the test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective major cardiac surgery under cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-05-17 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | Within 48 hours after surgery
  SCr was elevated ≥ 26.5 micromol/L or 1.5 times the baseline for SCr ≥ or urine output < 0.5 mL/kg/hour within 6 hours within 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University anesthesiology department, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No